CLINICAL TRIAL: NCT03565237
Title: Phase IV Multi-Center, Prospective, Interventional, Post-Marketing Study in Hemophilia B Patients in India Receiving RIXUBIS as On-demand or Prophylaxis Under Standard Clinical Practice
Brief Title: RIXUBIS PMS India (RIXUBIS PMS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 251602
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All Study Participants (Experimental): Study participants with Hemophilia B in India receiving Rixubis
  Interventions: Biological: RIXUBIS: On-Demand; Biological: RIXUBIS: Prophylaxis

INTERVENTIONS:
Biological: RIXUBIS: On-Demand — RIXUBIS used under standard clinical practice in India: On-Demand treatment.
  Other Names: BAX326; Recombinant Factor IX; rFIX; Coagulation Factor IX [Recombinant]; rFactor IX; BAX 326
Biological: RIXUBIS: Prophylaxis — RIXUBIS used under standard clinical practice in India: Prophylaxis treatment.
  Other Names: BAX326; Recombinant Factor IX; rFIX; Coagulation Factor IX [Recombinant]; rFactor IX; BAX 326

SUMMARY:
The purpose of this study is to characterize the safety and describe the effectiveness of RIXUBIS in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria

1. The participant or legally authorized representative (in case of study participants <18 years of age) gave written informed consent to participate in the study.
2. Participant has hemophilia B.
3. Participant is defined as previously-treated patient (PTP):

   * Participant aged ≥ 6 years that has been previously treated with plasma-derived and/or recombinant factor IX (FIX) concentrate(s) for a minimum of 150 exposure days (EDs).
   * Participant aged < 6 years that has been previously treated with plasma-derived and/or recombinant FIX concentrate(s) for a minimum of 50 EDs.
4. Participant has no evidence of a history of FIX inhibitors.
5. Participant is human immunodeficiency virus negative (HIV-); or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm^3, as confirmed by central laboratory at screening.
6. Participant is hepatitis C virus negative (HCV-) by antibody or PCR testing (if positive, antibody titer will be confirmed by polymerase chain reaction (PCR)), as confirmed by central laboratory at screening; or HCV+ with chronic stable hepatitis.
7. The participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria

1. Participant has known hypersensitivity or presence of any contraindication to RIXUBIS or its excipients including hamster protein.
2. Participant has evidence of an ongoing or recent thrombotic disease, fibrinolysis or disseminated intravascular coagulation (DIC).
3. Participant has a history of FIX inhibitors with a titer ≥ 0.6 Bethesda Units (BU) (as determined by the Nijmegen modification of the Bethesda assay or the assay, employed in the respective local laboratory) at any time prior to screening.
4. Participant has a detectable FIX inhibitor at screening, with a titer ≥ 0.6 BU as determined by the Nijmegen modification of the Bethesda assay in the central laboratory.
5. Participant has severe chronic liver disease as evidenced by, but not limited to, any of the following: International Normalized Ratio (INR) > 1.4 hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices.
6. Participant has severe chronic hepatic dysfunction [eg, ≥ 5 times upper limit of normal alanine aminotransferase (ALT), as confirmed by central laboratory at screening, or a documented INR > 1.5].
7. Participant has severe renal impairment (serum creatinine > 2.0 mg/dL), as confirmed by central laboratory at screening.
8. Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia B.
9. Participant's platelet count is < 100,000/mL.
10. Participant has a clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant's safety or compliance.
11. Participant is currently receiving, or is scheduled to receive during the course of the study, an immunomodulating drug (eg, corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day, or α-interferon) other than antiretroviral chemotherapy.
12. Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
13. Participant is a family member or employee of the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Sahyadri Super Speciality Hospital, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc64db2bf003ab45e07

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 study sites in India from 07 December 2018 to 11 August 2021.
Pre-assignment Details: A total 31 participants were screened, of which 25 participants were enrolled and received RIXUBIS treatment regimen (either on-demand or prophylaxis) based on discretion of the physician choice under standard clinical practice. No participants were enrolled in the on-demand treatment of RIXUBIS. Hence, no data collection and analysis were done during on-demand treatment of this study.
Groups:
- RIXUBIS: Prophylaxis Treatment: Participants received intravenous bolus of RIXUBIS prophylaxis treatment at a maximum infusion rate of 10 milliliter (mL) per (/) minute based on discretion of the physician for up to 6 months as standard clinical practice.
Period: Overall Study
Arm/Group | RIXUBIS: Prophylaxis Treatment
Started | 25
Safety Analysis Set (SAS) | 25
Effectiveness Full Analysis Set (EFAS) | 25
Completed | 23
Not Completed | 2
Not completed — Non-compliance of Investigational Product | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: SAS included all enrolled participants having received RIXUBIS at any time during the study.
Groups:
- RIXUBIS: Prophylaxis Treatment: Participants received intravenous bolus of RIXUBIS prophylaxis treatment at a maximum infusion rate of 10 mL/minute based on discretion of the physician for up to 6 months as standard clinical practice.
Arm/Group | RIXUBIS: Prophylaxis Treatment
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian: Indian | 24
  Race: More than one race | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Treatment-emergent Adverse Events (TEAEs) Related to RIXUBIS
Description: TEAE was defined as any event not presented prior to the initiation of the treatments or any event already present that worsens in either intensity or frequency following exposure to the treatments. A SAE was defined as any untoward medical occurrence that at any dose met one or more of the following criteria: outcome was fatal/resulted in death, life-threatening, required in-patient hospitalization or resulted in prolongation of an existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event that was not immediately life-threatening or resulted in death or required hospitalization but jeopardize the participant or required medical or surgical intervention to prevent any of the above outcomes. Relatedness to study drug was based on physician discretion. Number of participants with serious TEAEs related to RIXUBIS were reported.
Time Frame: From start of study drug administration up to End of treatment (EOT) (up to 6 months)
Population: SAS included all enrolled participants having received RIXUBIS at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | RIXUBIS: Prophylaxis Treatment
Number analyzed (Participants) | 25
Participants | 0

2. Secondary Outcome: Number of Participants With TEAEs Related to RIXUBIS
Description: TEAE was defined as any event not presented prior to the initiation of the treatments or any event already present that worsens in either intensity or frequency following exposure to the treatments. Relatedness to study drug was based on physician discretion. Number of participants with TEAEs related to RIXUBIS were reported.
Time Frame: From start of study drug administration up to EOT (up to 6 months)
Population: SAS included all enrolled participants having received RIXUBIS at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | RIXUBIS: Prophylaxis Treatment
Number analyzed (Participants) | 25
Participants | 0

3. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Clinical laboratory evaluations included clinical chemistry (biochemistry and endocrinology), hematology and urinalysis. Any change in clinical laboratory abnormalities which were deemed clinically significant by the investigator were recorded as TEAEs (defined as any event not presented prior to the initiation of the treatments or any event already present that worsens in either intensity or frequency following exposure to the treatments).
Time Frame: From start of study drug administration up to EOT (up to 6 months)
Population: SAS included all enrolled participants having received RIXUBIS at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | RIXUBIS: Prophylaxis Treatment
Number analyzed (Participants) | 25
Participants
  Hematology | 0
  Clinical chemistry | 0
  Urinalysis | 0

4. Secondary Outcome: Number of Participants Who Developed Binding Antibodies (Immunoglobulin G [IgG] and Immunoglobulin M [IgM]) to Factor IX (FIX)
Description: Binding antibodies (IgG and IgM) to FIX was determined using validated enzyme-linked immunosorbent assays (ELISAs) employing polyclonal anti-human IgG and IgM antibodies. Number of participants who developed binding antibodies (IgG and IgM) combined data to FIX were reported.
Time Frame: From start of study drug administration up to EOT (up to 6 months)
Population: SAS included all enrolled participants having received RIXUBIS at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | RIXUBIS: Prophylaxis Treatment
Number analyzed (Participants) | 25
Participants | 1

5. Secondary Outcome: Number of Participants Who Developed Binding Antibodies to Chinese Hamster Ovary (CHO) Proteins and rFurin
Description: Citrated plasma was assayed for the presence of antibodies to CHO protein and rFurin, derived from cultures of un-transfected cells. Testing for binding anti-CHO protein and rFurin antibodies was done on citrate-anti-coagulated plasma using an ELISA employing polyclonal anti-human IgG antibodies. Number of participants who developed binding antibodies to CHO proteins and rFurin were reported.
Time Frame: From start of study drug administration up to EOT (up to 6 months)
Population: SAS included all enrolled participants having received RIXUBIS at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | RIXUBIS: Prophylaxis Treatment
Number analyzed (Participants) | 25
Participants
  CHO Proteins | 0
  rFurin | 0

6. Secondary Outcome: Annualized Bleeding Rate (ABR) With Prophylactic Use of RIXUBIS
Description: The ABR was defined as the total number of unique bleeding episodes by participants reported during RIXUBIS treatment for prophylaxis, divided by the RIXUBIS treatment duration for prophylaxis and multiplied by 365.25. A bleeding episode was defined as subjective (pain consistent with a joint bleed) or objective evidence of bleeding which may or may not be associated to a trauma event (spontaneous bleeding). Bleeding occurring at multiple locations related to the same injury (e.g., knee and ankle bleed following a fall) was counted as a single bleeding episode.
Time Frame: From start of study drug administration up to EOT (up to 6 months)
Population: The EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | RIXUBIS: Prophylaxis Treatment
Number analyzed (Participants) | 23
episodes per participant per year | 0.914 (1.6896)

7. Secondary Outcome: Rate of Success of RIXUBIS for Treatment of Bleeding Episodes
Description: The success of RIXUBIS for treatment of bleeding episodes was defined by grouping the categories of "Excellent"/"Good" of the corresponding hemostatic effectiveness ratings of a 4 point Likert scale ("Excellent", "Good", "Moderate" and "None") by the participants/legally authorized representative (LAR) (participants less than (<) 12 years: LAR, participants greater than or equal to (>=) 12 years: self-assessment) for treatments given at home, or by the investigator for treatments given in the hospital/clinic. The rate of success of RIXUBIS for treatment of bleeding episodes was defined as: The number of successful bleeding episodes/total number of bleeding episodes where the treatment of the bleeding was rated *100. Rate of success of RIXUBIS for treatment of bleeding episodes, 95% confidence interval (CIs) was calculated using the exact Binomial CI (Clopper-Pearson method).
Time Frame: From screening up to EOT (up to 6 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | RIXUBIS: Prophylaxis Treatment
Number analyzed (Participants) | 6
Number analyzed (Bleeding episodes) | 6
percentage of bleeding episodes | 100 [54.1 to 100.0]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to EOT (up to 6 months)
Description: SAS included all enrolled participants having received RIXUBIS at any time during the study.
Arm/Group | RIXUBIS: Prophylaxis Treatment
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIXUBIS: Prophylaxis Treatment (N=25)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
No participants were enrolled in the on-demand treatment of RIXUBIS. Hence, no data collection and analysis was done during on-demand treatment of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT03565237/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT03565237/SAP_001.pdf